CLINICAL TRIAL: NCT04626011
Title: Impact of Total Teeth Extraction on Inflammation Marker's Levels in Patients Who Undergoing Cardiac Surgery: Clinical Trial.
Brief Title: Impact of Teeth Extraction on Inflammation Marker's Levels in Patients Who Undergoing Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, Bevilacqua Lorenzo, Clinical professor, DDS, MsC, University of Trieste
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BLorenzo
Record Dates: First submitted 2020-10-05; First posted 2020-11-12 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Inflammation Gum; Cardiac Surgery
Keywords: Tooth Extractions; Inflammation Markers; Cardiac Surgery
MeSH Terms: conditions — Gingivitis | interventions — Tooth Extraction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group One (Active Comparator): Participants receiving full mouth disinfection and extractions in one stage.
  Interventions: Procedure: Tooth extractions
- Group Two (Active Comparator): Participants receiving full mouth disinfection at stage one and extractions at stage two after 7 days.
  Interventions: Procedure: Tooth extractions

INTERVENTIONS:
Procedure: Tooth extractions — After blood collection tests, Periodontal analysis, Orthopantomography and Anamnestic record each group will receive a full mouth disinfection and needed extractions.
  Other Names: Inflammation markers evaluation

SUMMARY:
The aim of this study is to examine effects of dental treatments, surgical (extractions) and non-surgical procedures (non-surgical periodontal therapy), on serum levels for PCR, WBCs and PCT in patients needing a dental remediation before undergoing cardiac surgery.

DETAILED DESCRIPTION:
Introduction. The association between periodontal disease and cardiovascular disease is already established. Chronic inflammation of periodontal tissues primes the release of inflammatory markers such as: PCR, IL-1, IL-6 and TNF alpha and also,an even more accurate marker, procalcitonin (PCT).

Aim. The aim of this study is to examine effects of dental treatments, surgical (extractions) and non-surgical procedures (non-surgical periodontal therapy), on serum levels for PCR, WBCs and PCT in patients needing a dental remediation before undergoing cardiac surgery.

Materials and methods. This study is designed to be a clinical trial. 38 patients will be recruited at the Cardiological Center at Cattinara Hospital (ASUITS) and they will be treated in Maxillofacial Surgery and Stomatology Clinic at Major Hospital (ASUITS). Inclusion criteria: adult age, consciousness and willingness to sign an informed consent, anamnestic history of cardiovascular disease, also needing cardiac surgery and dental reclamation, stage 3-4 grade B-C for periodontal disease diagnosed . Exclusion criteria: pregnancy, genetic dysmorphisms which have an impact on the periodontal health status (Down Syndrome), diabetes or immune system disorders, HIV, hardly smoking, blood disorders, urgent cardiac surgery or a too large dental remediation to be performed in just 2 dental sessions, patients who underwent dental treatments in the previous 2 months. At baseline, all patients will undergo blood tests (blood cell count, PCR, PCT and WBC count), periodontal analysis (FMPS, FMBS and PISA index recording), orthopantomography and anamnestic record. Afterwards they will be assigned, randomly following a 1:1 ratio to Gruppo1 (fullmouth disinfection therapy + extractions all in one session) or Gruppo2 (fullmouth disinfection therapy and after one week extractions). All patients will undergo blood chemistry tests (CPR, PCT, WBC) after 1, 7 and 14 days.

Statistical analysis. All data will be presented as a mean and standard deviation, unless another method will be specified. After the control of parametric data distribution we will proceed with the statistical analysis of the different biomarkers recorded over time by ANOVA for repeated measurements and by t-test between the different groups in the same time intervals.

ELIGIBILITY:
Inclusion Criteria:

* adult age, consciousness and willingness to sign an informed consent, anamnestic history of cardiovascular disease, also needing cardiac surgery and dental reclamation, stage 3-4 grade B-C for periodontal disease diagnosed

Exclusion Criteria:

* pregnancy, genetic dysmorphisms which have an impact on the periodontal health status (Down Syndrome), diabetes or immune system disorders, HIV, hardly smoking, blood disorders, urgent cardiac surgery or a too large dental remediation to be performed in just 2 dental sessions, patients who underwent dental treatments in the previous 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2022-10-05 (Estimated); Study Completion 2022-10-05 (Estimated)

PRIMARY OUTCOMES:
Dental protocol to be followed in patients undergoing cardiac surgery by measuring changes in serum inflammatory markers. | Changes from baseline of serum inflammatory markers after 1 day, 7 days and 14 days.
  To find out which dental procedures protocol to be used to reduce serum inflammation markers as TNF alfa, IL 6, CPR, WBC and PCT values in patient undergoing cardiac surgery using a sample of 38 patients.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Bevilacqua, DDS, Principal Investigator — Clinica Stomatologia, Piazza dell'Ospitale 1, Ospedale Maggiore 34125 Trieste Italia
Locations (1):
- Department of Medical Sciences, University of Trieste, Trieste, Italy, Trieste, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cotti E, Cairo F, Bassareo PP, Fonzar F, Venturi M, Landi L, Parolari A, Franco V, Fabiani C, Barili F, Di Lenarda A, Gulizia M, Borzi M, Campus G, Musumeci F, Mercuro G. Perioperative dental screening and treatment in patients undergoing cardio-thoracic surgery and interventional cardiovascular procedures. A consensus report based on RAND/UCLA methodology. Int J Cardiol. 2019 Oct 1;292:78-86. doi: 10.1016/j.ijcard.2019.06.041. Epub 2019 Jun 17. PMID 31262607
- [Background] Chapple ILC, Mealey BL, Van Dyke TE, Bartold PM, Dommisch H, Eickholz P, Geisinger ML, Genco RJ, Glogauer M, Goldstein M, Griffin TJ, Holmstrup P, Johnson GK, Kapila Y, Lang NP, Meyle J, Murakami S, Plemons J, Romito GA, Shapira L, Tatakis DN, Teughels W, Trombelli L, Walter C, Wimmer G, Xenoudi P, Yoshie H. Periodontal health and gingival diseases and conditions on an intact and a reduced periodontium: Consensus report of workgroup 1 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S74-S84. doi: 10.1002/JPER.17-0719. PMID 29926944
- [Background] D'Aiuto F, Nibali L, Mohamed-Ali V, Vallance P, Tonetti MS. Periodontal therapy: a novel non-drug-induced experimental model to study human inflammation. J Periodontal Res. 2004 Oct;39(5):294-9. doi: 10.1111/j.1600-0765.2004.00741.x. PMID 15324349
- [Background] Ebersole JL, Machen RL, Steffen MJ, Willmann DE. Systemic acute-phase reactants, C-reactive protein and haptoglobin, in adult periodontitis. Clin Exp Immunol. 1997 Feb;107(2):347-52. doi: 10.1111/j.1365-2249.1997.270-ce1162.x. PMID 9030874
- [Background] Tonetti MS, D'Aiuto F, Nibali L, Donald A, Storry C, Parkar M, Suvan J, Hingorani AD, Vallance P, Deanfield J. Treatment of periodontitis and endothelial function. N Engl J Med. 2007 Mar 1;356(9):911-20. doi: 10.1056/NEJMoa063186. PMID 17329698
- [Background] Loos BG, Craandijk J, Hoek FJ, Wertheim-van Dillen PM, van der Velden U. Elevation of systemic markers related to cardiovascular diseases in the peripheral blood of periodontitis patients. J Periodontol. 2000 Oct;71(10):1528-34. doi: 10.1902/jop.2000.71.10.1528. PMID 11063384